CLINICAL TRIAL: NCT05855369
Title: A Randomized Controlled Trial of Smell Training and Trigeminal Nerve Stimulation in the Treatment of COVID-related Persistent Smell Loss
Brief Title: Study of Chemosensory Enhancement Through Neuromodulation Training (SCENT for Long COVID)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Bernadette Cortese, Assistant Professor of Psychiatry and Behavioral Sciences, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00127790; R01DC021179 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-11 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Smell Dysfunction; Olfactory Disorder; Long COVID
Keywords: COVID-19; Parosmia; Hyposmia; Anosmia; Phantosmia; Dysosmia; Olfactory Training; Neuromodulation; Non-invasive Brain Stimulation
MeSH Terms: conditions — Olfaction Disorders; Post-Acute COVID-19 Syndrome; COVID-19; Anosmia | interventions — Transcutaneous Electric Nerve Stimulation; Olfactory Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A separate outcomes assessor, blind to treatment intervention for all participants, will perform all clinician-administered primary outcomes (i.e. olfactory function determined by Sniffin' Sticks, ratings for odor intensity/hedonics, clinician-administered assessment of cognitive function, and the clinical global impressions for smell dysfunction). This outcomes assessor will not be involved with any other aspects of the trial.
  Additionally, the participant will be blind to ST versus PBO group assignment, but not TNS+ST assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combination Trigeminal Nerve Stimulation (TNS) and active Smell Training (ST) (Active Comparator): 30 minutes of once/day TNS and twice/day ST conducted 5 days/week for 12 weeks and a total of 60 stimulation and 120 smell training sessions
  Interventions: Device: Trigeminal Nerve Stimulation (TNS); Other: Active Smell Training (ST)
- Active Smell Training (ST) (Active Comparator): 5 minutes of daily ST conducted twice/day, 5 days/week for 12 weeks and a total of 120 training session
  Interventions: Other: Active Smell Training (ST)
- Placebo Smell Training (PBO) (Placebo Comparator): 5 minutes of daily PBO conducted twice/day, 5 days/week for 12 weeks and a total of 120 training sessions
  Interventions: Other: Placebo Smell Training (PBO)

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation (TNS) — Non-invasive, pain-free, low-level electrical stimulation to the forehead to modulate the trigeminal nerve and enhance smell function through activation of the highly connected olfactory-intranasal trigeminal brain circuits.
  Other Names: Transcutaneous Electrical Nerve Stimulation
  Arms: Combination Trigeminal Nerve Stimulation (TNS) and active Smell Training (ST)
Other: Active Smell Training (ST) — Sniffing various higher intensity odorant chemicals while performing odor-related cognitive tasks. 16 odorant chemicals will be used for training including: 2 phenyl ethanol, eugenol, lemon, eucalyptus, cinnamon, peppermint, coffee, mandarin, lavender, vanilla, lilac, ginger, chocolate, thyme, banana, and bacon.
  Other Names: Olfactory Training
  Arms: Active Smell Training (ST); Combination Trigeminal Nerve Stimulation (TNS) and active Smell Training (ST)
Other: Placebo Smell Training (PBO) — Sniffing the same lower intensity odorant chemicals (i.e. N-butanol and 2-phenyl ethanol) over the course of the trial and performing no odor-related cognitive tasks.
  Arms: Placebo Smell Training (PBO)

SUMMARY:
Persistent smell loss that can include diminished or distorted smell function is a common symptom of long COVID syndrome. There are limited treatment options for long COVID-related smell loss. This study aims to determine the efficacy of two at-home treatments, smell training and non-invasive trigeminal nerve stimulation. This study requires participants to conduct daily at-home treatment sessions, attend three in-person study visits at the MUSC Department of Psychiatry and Behavioral Sciences, and complete electronic questionnaires over the 12-week trial, and again at the six-month timepoint. Participants in this trial may benefit directly with an improvement in sense of smell. However, participation may also help society more generally, as this study will provide new information about long COVID-related smell loss and its treatment.

DETAILED DESCRIPTION:
Sudden smell loss (SL), a hallmark feature of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-coV-2/COVID), frequently persists well past the initial recovery; rates of unresolved anosmia (total loss) are 21%, with unresolved hyposmia (reduced smell) or parosmia (distorted smell) higher at nearly 50%. SL is now recognized as a core symptom of "long COVID" (LC), which also includes other impairments in mood, cognition, and sleep. Given that SL itself can negatively impact many of the same problems being recognized in the symptomatology of LC, it is likely that SL is both a symptom of LC and a contributing factor that worsens other LC symptoms (i.e. mood, cognition, sleep, etc.). As such, successful treatment of SL could also help to improve these other LC symptoms.

Smell/olfactory training (ST) is currently being studied as a treatment for COVID-related SL. Classic ST requires twice daily practice of sniffing odorants over the course of 3 months to regenerate olfactory neurons, engage smell-related cognitive functions, and retrain the brain to smell. ST is promising as a stand-alone treatment. However, its limitations include the burden of many months of daily practice that often leads to sub-optimal compliance and dropout.

The current study aims to determine whether the benefits of ST can be accelerated and enhanced by using a novel, adjunct neuromodulatory intervention to conventional ST. Trigeminal nerve stimulation (TNS) is a non-invasive, pain-free, method of neuromodulation that delivers low levels of electrical stimulation to the trigeminal circuit, having potential to enhance smell function through activation of the highly connected olfactory-intranasal trigeminal systems. Prior work demonstrated TNS-enhanced psychophysical detection of odorants. Yet the effects of TNS are extensive, i.e. improved executive functioning (e.g. attention), sleep quality, and daytime sleepiness, as well as therapeutic efficacy across a number of neuropsychiatric disorders. Thus, TNS-as an adjunct to ST-may not only improve overall efficacy and speed of recovery of SL, but may help to treat some of the other symptoms of LC that ST, and improvement in smell function, may not fully resolve.

This randomized, controlled trial (RCT) of ST and combination TNS and ST in adults with COVID-related SL will use a 3- group design: Group 1) Active ST (N=60), Group 2) Placebo ST (PBO, N=60), and Group 3) Active TNS plus Active ST (N=60). Our primary objectives are to 1) determine the efficacy of ST versus potential natural gains in function, 2) determine the TNS-enhanced effects of ST on SL, and 3) determine whether TNS+ST is more efficacious than ST in treating the other symptoms of LC.

ELIGIBILITY:
Inclusion Criteria:

* treatment-seeking for COVID-related persistent SL (anosmia, hyposmia, phantosmia or parosmia)
* at least 1-month from SARS-coV-2 PCR-positive and/or rapid home-positive tests
* normal sense of smell prior to COVID
* naïve to both smell training (ST) and trigeminal nerve stimulation (TNS)
* able to comprehend English and provide informed consent

Exclusion Criteria:

* history of head injury (e.g. sport, accident, combat blast)
* sinonasal condition (e.g. upper respiratory infection, rhinosinusitis, polyps)
* neurological disorder (e.g. epilepsy, neurodegenerative disorder, narcolepsy)
* serious mental illness (e.g. schizophrenia, bipolar, or other psychotic disorder)
* suicidal ideation within the last month
* current (≤6 months) heavy cigarette smoker (heavy defined as ≥ 10 pack-years)
* oral/nasal steroids or other intranasal medications within the last month
* immunomodulatory medications
* pregnant or trying to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Psychophysical Olfactory Function from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  Sniffin' Sticks (Bughardt Messtechnik, Wedel Germany) will be used to determine odor threshold (T), odor discrimination (D), and odor identification (I), each on 16-point scales, and summed for a total TDI score. Higher scores indicate better function.
Change in Perceived Intensity of Odorants from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  Perceived intensity on 100-mm visual analog scales with anchor points: 0="imperceptible" to 100="extremely intense" will be rated for suprathreshold concentrations of PEA, vanilla, eugenol, and eucalyptus.
Change in Perceived Hedonics of Odorants from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  Perceived hedonics on 100-mm visual analog scales with anchor points: 0="extremely unpleasant" to 100="extremely pleasant".
Change in Olfactory-related Quality of Life from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Modified Questionnaire of Olfactory Disorders-Negative Statements (QOD-NS) consists of 17 negative statements (rated on a scale from 0 to 3; total score ranging from 0 to 51), with lower scores indicating better olfactory-related quality of life.
Change in Impact of Olfactory Loss from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Impact of Olfactory Loss Visual Analog Scale (IOL-VAS) consists of 9 separate items assessing the impact of olfactory loss upon mood, food enjoyment, social interactions, safety, hygiene, sex, cooking, appetite, and weight changes, rated from 0 (no impact) to 10 (biggest impact possible).

SECONDARY OUTCOMES:
Change in Long COVID Symptoms from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  53 long COVID symptoms (scored from 0-53 reflecting the number of different symptoms experienced) and the impact of those symptoms (scored from 0=no impact to 10=maximal impact) will be obtained.
Change in Sustained Attention from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Sustained Attention to Response Task (SART) is a computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target (often the digit 3) presented amongst a background of frequent non-targets (0-2, 4-9).
Change in Cognitive Function from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The NIH Toolbox Cognitive Battery is a widely used assessment for detecting cognitive impairment. This test assesses short-term memory, executable performance, attention, and focus.
Change in Mood State from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Profile of Mood States Short Form (POMS-SF) is a psychological rating scale used to assess transient, distinct mood states across six different dimensions including Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, and Confusion or Bewilderment.
Change in Sleep Quality from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. Scores greater than 5 are indicative of a sleep disturbance.
Change in Excessive Daytime Sleepiness from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Epworth Sleepiness Scale (ESS) is a measure intended to assess daytime sleepiness. Items consist of 8 different activities which are rated according to how likely it would be to doze off or fall asleep if engaged in that activity. A score of 10 or more is indicative excessive daytime sleepiness.
Change in Symptoms of Depression from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a self-administered 9-item questionnaire to screen for the presence and severity of depression. Items are rated on a 3pt scale ranging from 0="Not at all" to 3="Nearly every day". Total score ranges from 0-27 and is used to classify depression severity: 0-4=None/Minimal; 5-9=Mild; 10-14=Moderate; 15-19=Moderately Severe; 20-27=Severe.
Change in Symptoms of Anxiety from Baseline to 4 and 12 Weeks | 2 times: 4 weeks, 12 weeks
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item questionnaire to screen for presence and severity of anxiety disorder. Items are rated on a 3pt scale ranging from 0="Not at all" to 3="Nearly every day". Total score ranges from 0 to 21 and is used to classify anxiety severity: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), 15-21 (severe anxiety).

OTHER OUTCOMES:
Treatment Feasibility, Acceptability, and Fidelity at 4 and 12 weeks | 2 times: 4 weeks, 12 weeks
  Quantitative measurements will include the number of 1) sessions completed (completion rate), 2) technical problems, 3) adverse events, 4) study drop-out, and 5) the number of study-issued treatment cases returned at the end of treatment. The Feasibility of Intervention Measure (FIM) and the Acceptability of Intervention Measure (AIM) will be used. Both the FIM and AIM contain 4 items that are scored on a 5-point scale (1=completely disagree to 5=completely agree). Responses are averaged across the 4 items, with a score of 4 or more indicating adequate feasibility and acceptability of an intervention. Fidelity (i.e. adherence) that the treatment is delivered as intended will be measured by study staff who will rate adherence on a 5-point scale (1=little to 5=complete). Qualitative data using open-ended questions regarding the nature of any technical problems and the reasons for missed treatment sessions will be assessed.
Durability of Treatment on Subjective Olfactory Function at the 6-month Follow Up | 1 time: 6 months
  Subjective function will be assessed with the QOD-NS and IOL-VAS.
Durability of Treatment on Long COVID Symptoms at the 6-month Follow Up | 1 time: 6 months
  53 long COVID symptoms (scored from 0-53 reflecting the number of different symptoms experienced) and the impact of those symptoms (scored from 0=no impact to 10=maximal impact) will be obtained.
Durability of Treatment on Mood at the 6-month Follow Up | 1 time: 6 months
  Mood will be assessed with the PHQ-9, GAD-7, and POMS-SF
Durability of Treatment on Sleepiness and Sleep Quality at the 6-month Follow Up | 1 time: 6 months
  Sleepiness and Sleep Quality will be assessed with the ESS and PSQI

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Original data (de-identified) will be available to other researchers upon request. Human subjects' rights to privacy will be protected and the identity of human subjects will not be revealed with any request.
Supporting Information: Study Protocol
Time Frame: IPD will be shared after the primary data analyses are complete and our final findings are published.
Access Criteria: Information on where the data will be available and how to access it will be published with all publications/presentations that come from this study